CLINICAL TRIAL: NCT03163784
Title: SHIFT: Studying HIV Immunology After Fecal Transplant
Acronym: SHIFT
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study closed because of shifting research priorities and interests.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, DOUGLAS KWON, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2016P002317
Record Dates: First submitted 2017-05-18; First posted 2017-05-23 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: HIV/AIDS; Dysbiosis; Inflammation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Dysbiosis; Inflammation | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Placebo Comparator): Weekly placebo (for Fecal Inoculum Capsule) treatment with placebo pre-treatment.
  Interventions: Biological: Placebo (for Fecal Inoculum Capsule); Drug: Antibiotic Placebo
- Arm B (Experimental): Weekly Fecal Inoculum Capsule treatment with placebo pre-treatment.
  Interventions: Biological: Fecal Inoculum Capsule; Drug: Antibiotic Placebo
- Arm C (Experimental): Weekly Fecal Inoculum Capsule treatment with antibiotic pre-treatment.
  Interventions: Biological: Fecal Inoculum Capsule; Drug: Antibiotic

INTERVENTIONS:
Biological: Fecal Inoculum Capsule — Sieved fecal matter prepared in glycerol/saline solution
  Arms: Arm B; Arm C
Biological: Placebo (for Fecal Inoculum Capsule) — Placebo capsule manufactured to mimic Fecal Inoculum Capsules
  Other Names: Placebo
  Arms: Arm A
Drug: Antibiotic — Antibiotic pre-treatment
  Arms: Arm C
Drug: Antibiotic Placebo — Placebo tablets manufactured to mimic antibiotics
  Arms: Arm A; Arm B

SUMMARY:
SHIFT is a randomized, longitudinal, prospective, blinded, three-arm study to determine the safety and tolerability of Fecal Microbiota Transplant (FMT) in HIV-infected participants on stable antiretroviral therapy (ART).

DETAILED DESCRIPTION:
This study is designed to test the safety and tolerability of Fecal Microbiota Transplant (FMT) in HIV infected individuals on stable antiretroviral therapy (ART). Additionally, the study will examine potential effects of FMT on HIV immune activation, which has been linked to HIV disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 18 - 75 years.
2. HIV-1 positive:
3. Ability and willingness of participant or legal guardian/representative to provide informed consent.

Exclusion Criteria:

1. Patients with a history of significant allergy to tree nuts, peanuts, shellfish, and/or eggs, vancomycin, levofloxacin, or metronidazole, chocolate/cocoa or gelatin; or unwillingness to ingest gelatin (in placebo capsules)
2. Use of investigational therapies or investigational vaccines within 90 days prior to study entry
3. Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to entry
4. History of positive HCV antibody with detectable HCV RNA in plasma within 48 weeks prior to study entry.
5. History of positive HBsAg within 48 weeks prior to study entry
6. Liver cirrhosis, history of C. difficile infection, history of inflammatory bowel disease, bariatric surgery, total colectomy, colon or rectal anastomosis, bowel resection, or current colostomy.
7. Current diagnosis of diabetes
8. BMI >35
9. Either breastfeeding or pregnant within 24 weeks prior to study entry
10. Tendinopathy or peripheral neuropathy (potentially exacerbated by antibiotic pretreatment)
11. Use of immunosuppressives, immune modulators, or antineoplastic agents for more than 3 consecutive days within the 60 days prior to study entry.
12. Use of probiotics and prebiotics (supplements and products) within 30 days of the study. Yogurt with live cultures is allowed.
13. Diagnosed bacterial enteric infection within 30 days prior to study entry.
14. Acute diarrhea within 30 days of study entry.
15. Weight loss or gain of more than 25 pounds in the 24 weeks prior to study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
FMT-related adverse events | 30 weeks
  Safety of FMT in stably suppressed HIV infected recipients on ART

SECONDARY OUTCOMES:
Immune and metabolic markers | 30 weeks
  Changes in immune and metabolic markers such as CD4 T cell activation and sCD14 levels.
Microbiome structure | 30 weeks
  Identify and characterize how FMT alters enteric microbiome structure.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Kwon, MD, PhD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: Undecided